CLINICAL TRIAL: NCT00005985
Title: Primed Peripheral Blood Stem Cell Autologous Transplantation for Lymphoma and Hodgkin's Disease
Brief Title: Filgrastim and Chemotherapy Followed by Peripheral Stem Cell Transplant in Treating Patients With Hodgkin's Lymphoma or Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: 1996LS155; UMN-MT-9527; UMN-MT-1995-27
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Lymphoma
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I adult Burkitt lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage I adult T-cell leukemia/lymphoma; stage II adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; contiguous stage II small lymphocytic lymphoma; noncontiguous stage II small lymphocytic lymphoma; recurrent small lymphocytic lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Filgrastim; Carmustine; Cyclophosphamide; Cytarabine; Dexamethasone; Etoposide; Mitoxantrone; Peripheral Blood Stem Cell Transplantation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: filgrastim
Drug: carmustine
Drug: cyclophosphamide
Drug: cytarabine
Drug: dexamethasone
Drug: etoposide
Drug: mitoxantrone hydrochloride
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplant may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells. Colony-stimulating factors such as filgrastim may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of chemotherapy.

PURPOSE: This phase II trial is studying how well giving filgrastim together with chemotherapy and peripheral stem cell transplant works in treating patients with Hodgkin's lymphoma or non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the clinical outcomes, survival, and morbidity of transplantation in patients with Hodgkin's lymphoma or non-Hodgkin's lymphoma when treated with filgrastim (G-CSF) followed by high dose chemotherapy plus G-CSF followed by autologous peripheral blood stem cell (PBSC) transplantation.
* Determine whether sufficient PBSC can be collected for use in autologous transplantation in these patients when mobilized with hematopoietic growth factor alone compared to chemotherapy plus growth factor.
* Determine whether these primed PBSC support prompt lymphoid and myeloid hematopoietic recovery after transplantation in these patients.
* Compare the numbers of committed progenitor cells and/or primitive, pluripotential hematopoietic stem cells with these two priming techniques.
* Compare the numbers of tumor cells in cryopreserved PBSC following these priming techniques.
* Evaluate response and extended relapse free survival in conjunction with rapid hematopoietic reconstitution and limited transplant associated morbidity and mortality in these patients when treated with these regimens.

OUTLINE: In the first priming phase, patients receive filgrastim (G-CSF) subcutaneously (SQ) daily on days 1-7 and peripheral blood stem cells are collected on days 6-8.

At least 48 hours after the last dose of G-CSF and after the third leukapheresis, patients receive the second priming, which consists of cyclophosphamide IV over 2 hours on day 1 and cytarabine IV over 1 hour every 12 hours for a total of 2 doses on day 1. Patients also receive mitoxantrone IV over 1 hour daily and dexamethasone IV every 12 hours for a total of 4 doses on days 1-2. Patients receive G-CSF SQ daily beginning on day 4 and continuing until the completion of leukapheresis. PBSC are collected on 3 consecutive days after blood counts recover.

In the transplant phase, patients with non-Hodgkin's lymphoma who have not exceeded pretransplant radiotherapy limits receive cyclophosphamide IV over 2 hours on days -7 and -6 and total body irradiation twice daily on days -4 through -1. Autologous PBSC are reinfused on day 0. Patients receive G-CSF IV daily beginning on day 0 and continuing until day 21 or until blood counts recover.

Patients with Hodgkin's lymphoma or patients with non-Hodgkin's lymphoma who have exceeded pretransplant radiotherapy limits receive cyclophosphamide IV over 2 hours daily on days -6 through -3, carmustine IV over 1 hour on day -6, and etoposide IV over 4 hours every 12 hours for a total of 6 doses on days -6 through -4. Autologous PBSC are reinfused on day 0. Patients also receive G-CSF IV daily beginning on day 0 and continuing until day 21 or until blood counts recover.

All patients receive radiotherapy for any residual nodal masses measuring at least 2 cm 5 days a week beginning on day 28.

Patients are followed at day 100, then every 3 months for 1 year, then every 6 months for 2 years, and then annually thereafter.

This was changed to a treatment guideline study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* One of the following histologically confirmed diagnoses

  * High grade non-Hodgkin's lymphoma:

    * Immunoblastic or small noncleaved cell lymphoma (Burkitt's or non-Burkitt's) in complete or partial remission after initial therapy
    * Localized (stage I or Zeigler stage A) small noncleaved (Burkitt's or non-Burkitt's) after relapse or incomplete response to initial therapy
    * Lymphoblastic lymphoma in second or greater complete or partial response
    * High risk lymphoblastic lymphoma in first complete remission or after initial therapy (high risk factors include stage IV disease, LDH greater than 2 times normal, and 2 or more extranodal sites)
  * Intermediate grade non-Hodgkin's lymphoma:

    * Diffuse large cell lymphoma
    * Diffuse mixed cell lymphoma
    * Diffuse small cleaved cell lymphoma
    * Follicular large cell lymphoma
    * In second or greater complete or partial remission OR
    * High risk in first complete remission or after initial therapy

      * High risk features include:

        * No complete response after 12 weeks of initial combination chemotherapy
        * Bulky disease (greater than 10 cm nodal masses or mediastinal disease involving greater than 1/3 of the chest diameter
        * Malignant pleural effusion
        * Liver involvement
        * LDH greater than 2 times upper limit of normal at diagnosis
        * At least 2 extranodal sites
  * Low grade non-Hodgkin's lymphoma:

    * Follicular small cleaved cell lymphoma
    * Follicular mixed cell lymphoma
    * Diffuse small lymphocytic lymphoma
    * In first or greater complete response OR
    * Following initial treatment if complete response is not achieved
    * In second or greater complete or partial response if treated at diagnosis without clinical symptoms necessitating treatment
  * T-cell lymphoma (nonlymphoblastic, intermediate, or high grade lymphomas) after initial therapy whether or not complete response is achieved
  * Hodgkin's lymphoma

    * Stage I and II disease treated with primary radiotherapy and failure of at least one combination chemotherapy regimen
    * Stage III and IV disease with failure on mechlorethamine, vincristine, procarbazine, and prednisone (MOPP)-like regimen, alternative noncross resistant regimen (e.g., doxorubicin, bleomycin, vinblastine, and dacarbazine [ABVD]), or a combination (e.g., MOPP-ABV)
    * High risk features allowed including:

      * Failure to achieve initial complete remission with MOPP and/or ABVD and crossover or hybrid therapy
      * Relapse within 6 months after initial therapy
      * Relapse after initial radiotherapy with complete response longer than 1 year since initial therapy and subsequent failure on MOPP and/or ABVD or hybrid
    * Bulky mediastinal disease after initial therapy and residual mass of at least 5 cm with other features of persisting disease (e.g., Gallium scan positive, high LDH, enlarging on serial x-rays, or positive biopsy)
* No HIV or HTLV-1 associated lymphomas
* No resistant or refractory lymphoma (no partial response following up to 3 courses of combination chemotherapy)
* No active ischemic or degenerative CNS disease NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age:

* 70 and under

Performance status:

* Age 65-70 years:

  * Karnofsky 80-100%
* Under 65 years:

  * ECOG 0-1 (2 allowed if symptoms are directly related to lymphoma)

Life expectancy:

* Greater than 8 weeks

Hematopoietic:

* Not specified

Hepatic:

* No prior or current chronic liver disease
* Bilirubin no greater than 1.5 mg/dL
* AST and alkaline phosphatase less than 2 times normal

Renal:

* Age 65-70 years:

  * Creatinine clearance greater than 60 mL/min (if creatinine at least 1.5 mg/dL)
* Under 65 years:

  * Creatinine no greater than 1.5 mg/dL OR
  * Creatinine clearance greater than 50 mL/min

Cardiovascular:

* LVEF at least 45% by MUGA
* No symptoms of cardiac disease
* No active ischemic heart disease
* No uncontrolled hypertension

Pulmonary:

* Age 65-70 years:

  * If history of smoking or respiratory symptoms, spirometry and DLCO must be greater than 50% of predicted
* All ages:

  * No obstructive airway disease
  * No resting hypoxemia (PO_2 less than 80)
  * DLCO at least 50% of predicted

Other:

* No poorly controlled diabetes

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* Must have prior chemotherapy to attempt to achieve complete response

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* No radiotherapy to residual disease prior to transplantation

Surgery:

* Not specified

Other:

* Concurrent IV antibiotic therapy allowed for fever or signs of infection

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2000-08; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Disease-free survival at 2 years

SECONDARY OUTCOMES:
Relapse or progression transplant related mortality at 1½ years

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J. Weisdorf, MD, Study Chair — Masonic Cancer Center, University of Minnesota
Locations (1):
- University of Minnesota Cancer Center, Minneapolis, Minnesota, United States